CLINICAL TRIAL: NCT04939701
Title: A Phase 1/2 Open-label Study Investigating the Safety, Tolerability and Efficacy of ASP0739 as a Single Agent and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors Known to Express NY-ESO-1
Brief Title: Study of ASP0739 Alone and With Pembrolizumab in Advanced Solid Tumors With NY-ESO-1 Expression Participants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The comprehensive assessment of other studies indicated the lack of significant monotherapy activity, therefore, team decided to terminate the study.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0739-CL-0101
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; NSCLC; ESCC; Solid Tumors
Keywords: NY-ESO-1; ASP0739; Solid Tumor; NSCLC; ESCC; MRCL; Ovarian Cancer; R/R SS
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Phase 1): ASP0739 1x10^7 cells/mL (Experimental): Participants with Relapsed/Refractory (R/R) solid tumors known to express New York esophageal squamous cell carcinoma 1 (NY-ESO-1) received intravenous (IV) infusion of ASP0739 (human embryonic kidney cell [HEK293] transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^7 cells/milliliters (mL) at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a partial response (PR) or stable disease (SD) (1 cycle= 28 days). .
  Interventions: Drug: ASP0739
- Dose Escalation (Phase 1): ASP0739 1x10^8 cells/mL (Experimental): Participants with R/R solid tumors known to express NY-ESO-1 received IV infusion of ASP0739 (HEK293 transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a PR or SD (1 cycle= 28 days).
  Interventions: Drug: ASP0739
- Dose Expansion (Phase 2): ASP0739 1x10^8 cells/mL (Experimental): Participants with synovial sarcoma (SS), myxoid/round cell liposarcoma (MRCL), ovarian cancer and other solid tumors known to express NY-ESO-1 (melanoma, non-small cell lung cancer [NSCLC] adenocarcinoma and squamous cell and esophageal squamous cell carcinoma [ESCC]) received IV infusion of ASP0739 (HEK293 transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a PR or SD (1 cycle= 28 days).
  Interventions: Drug: ASP0739

INTERVENTIONS:
Drug: ASP0739 — Intravenous (IV)

SUMMARY:
The purpose of this study was to evaluate the safety, and tolerability of ASP0739, when administered as a single agent and in combination with pembrolizumab.

This study also evaluated the clinical response and other measures of anticancer activity of ASP0739 when administered as a single agent and in combination with pembrolizumab based on central and local assessment.

DETAILED DESCRIPTION:
The study comprised of 2 phases. Phase 1 (dose escalation) included participants with solid tumors known to express New York esophageal squamous cell carcinoma 1 (NY-ESO-1). Phase 2 (ASP0739 as single agent and in combination with pembrolizumab) included participants with relapsed/refractory Synovial Sarcoma (SS), myxoid/round cell liposarcoma (MRCL), and ovarian cancer who had not responded to Standard of Care (SOC) or were ineligible for standard therapy. Phase 2 single agent also included a cohort of participants with select solid tumors known to express NY-ESO-1 (melanoma, Non Small Cell Lung Cancer-adenocarcinoma [NSCLC], squamous cell and esophageal squamous cell carcinoma [ESCC]). Japanese participants were only enrolled into the monotherapy arm of the dose expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Dose Escalation only:

- Participant has relapsed/refractory (R/R) solid tumor known to express NY-ESO-1 after completing available Standard of Care (SOC) therapy or is not a candidate for SOC therapy. NY-ESO-1 expression status is not required for participant entry.

Safety Lead-in, Phase 2 Single agent and Combination Therapy only:

* Participant has relapsed/refractory (R/R) synovial sarcoma (SS) or myxoid/round cell liposarcoma (MRCL) disease after undergoing available SOC treatment or is not a candidate for SOC therapy (must have previously received either an anthracycline or ifosfamide containing regimen or another systemic regimen, if not a candidate for either agent).

  * Participant has not received prior checkpoint inhibitor therapy (i.e., Programmed Cell Death Protein 1 [PD-1]/Programmed Death Ligand 1 [PD-L1] treatment naive)
  * SS: confirmation by the presence of a translocation between SYT on the X chromosome and SSX1, SSX2, or SSX4 on chromosome 18 (may be presented in the pathology report as t [X;18]).
  * MRCL: confirmation by the presence of the reciprocal chromosomal translocation t (12;16) (q13;p11) or t(12;22)(q13;q12).
* Participant has R/R ovarian cancer that is:

  * platinum resistant OR platinum-sensitive, but the participant is not a candidate for platinum or other SOC therapy.
  * Participant has not received prior checkpoint inhibitor therapy (i.e., naive PD-1/PD-L1 treatment participants).
* Participant has R/R solid tumor (melanoma, non-small cell lung cancer [NSCLC]-adenocarcinoma and squamous cell, or esophageal squamous cell carcinoma [ESCC]) after available SOC treatment or is not a candidate for SOC therapy (single-agent only).
* Participant consents to provide an archival tumor specimen in a tissue block or unstained serial slides prior to IP administration.
* Participant in phase 2 consents to provide tumor specimen obtained within 56 days prior to first dose of study treatment, as tissue block or unstained serial slides.
* Participant in phase 2 consents to undergoing a tumor biopsy (core needle biopsy or excision) during the treatment period.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of <= 2.
* Participant with life expectancy of >= 12 weeks at the time of screening.
* Participant must meet criteria for clinical laboratory tests during screening period.
* A female participant is eligible to participate if she is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final investigational product (IP) administration.
* Female participant must not be breastfeeding at screening or during the study period and for 6 months after the final IP administration.
* Female participant must not donate ova at screening and throughout the study period and for 6 months after the final IP administration.
* A male participant with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 6 months after the final IP administration.
* Male participant must not donate sperm starting at screening and throughout the study period and for 6 months after the final IP administration.
* Participant agrees not to participate in another interventional study while on treatment.
* Participant measurable disease according to RECIST 1.1. For participant with only 1 measurable lesion and prior radiotherapy, the lesion must be outside the field of prior radiotherapy or must have documented progression following radiation therapy.

Exclusion Criteria:

* Participant has persistent non-hematological toxicities of >= grade 2 (National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0), with symptoms and objective findings from treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation or surgery).
* Participant has received any of the following therapies (for inclusion in the study, all abnormalities must have returned to <= grade 1):

  * Systemic immunomodulators (checkpoint inhibitors)-except the dose escalation phase and the NY-ESO-1 solid tumor (melanoma, NSCLC-adenocarcinoma and squamous cell and ESCC) cohorts in the dose expansion phase of monotherapy, which may have received prior checkpoint inhibitor therapy
  * Immunosuppressive drugs including steroids <= 14 days prior to treatment
  * Cytotoxic agents <= 14 days prior to treatment
  * Investigational agent <= 21 days prior to treatment or 5 half-lives, whichever is shorter
  * Radiation therapy <= 21 days prior to treatment
* Participant has clinically active or untreated nervous system metastases. Participants with previously treated Central Nervous System (CNS) metastases are eligible, if they are clinically stable and have no evidence of CNS progression by imaging for at least 4 weeks prior to start of study treatment and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone or > 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Participant has an active autoimmune disease. Participant with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy, or skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment are allowed.
* Participant was discontinued from prior immunomodulatory therapy due to a grade >= 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Participant has known history of serious hypersensitivity reaction to a known ingredient of ASP0739 or pembrolizumab or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Participant has a prior malignancy active (i.e., requiring treatment or intervention) within the previous 2 years prior to screening visit, except for locally curable malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
* Participant has received a prior allogeneic bone marrow or solid organ transplant.
* Participant has an active uncontrolled infection within 14 days of treatment.
* Participant is known to have human immunodeficiency virus infection.
* Participant has active hepatitis B or C or other active hepatic disorder or participant is on hepatitis treatment. Hepatitis C RNA testing is not required in participants with negative hepatitis C antibody testing.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has had a major surgical procedure and has not completely recovered within 28 days prior to the start of study treatment.
* Participant has had a myocardial infarction or unstable angina within 6 months prior to the start of study treatment or currently has an uncontrolled illness including, but not limited to, symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant is expected to require another form of anti-cancer therapy while on study treatment.
* Participant has a known or suspected hypersensitivity to bovine-derived protein or has suspected hypersensitivity to any ingredients of ASP0739.

Additional Exclusion Criteria for Participants in Combination Therapy Cohorts

* Participants with a history of myocarditis or congestive heart failure (as defined by New York Heart Associated Functional Classification III or IV), as well as unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry.
* Participants with active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids.
* Participants with baseline pulse oximetry < 92% "on Room air."
* Participants must not have known microsatellite instability-high or deficient MisMatch Repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - University of Miami, Miami, Florida
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - NYU Perlmutter Cancer Center, New York, New York
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/0739-CL-0101/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14599&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Relapsed/Refractory (R/R) solid tumors and with synovial sarcoma (SS), myxoid/round cell liposarcoma (MRCL), ovarian cancer and other solid tumors known to express New York esophageal squamous cell carcinoma 1 (NY-ESO-1) (melanoma, non-small cell lung cancer [NSCLC] adenocarcinoma and squamous cell and esophageal squamous cell carcinoma [ESCC]) were recruited.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study. Study was terminated at dose expansion monotherapy after the comprehensive assessment of other studies that indicated the lack of sufficient monotherapy activity, therefore, team decided to terminate the study.
Groups:
- Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL: Participants with R/R solid tumors known to express NY-ESO-1 received intravenous (IV) infusion of ASP0739 (human embryonic kidney cell [HEK293] transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^7 cells/milliliters (mL) at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a partial response (PR) or stable disease (SD) (1 cycle= 28 days).
- Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL: Participants with SS, MRCL, ovarian cancer and other solid tumors known to express NY-ESO-1 (melanoma, NSCLC adenocarcinoma and squamous cell and ESCC) received IV infusion of ASP0739 (HEK293 transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a PR or SD (1 cycle= 28 days).
Period: Phase 1: Dose Escalation (168 Days)
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Started | 4 | 7 | 0
Completed | 1 | 0 | 0
Not Completed | 3 | 7 | 0
Not completed — Progressive disease | 0 | 5 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Phase 2: Dose Expansion (168 Days)
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Started | 0 | 0 | 5
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 4
Not completed — Progressive disease | 0 | 0 | 3
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF). All participants who took at least 1 dose of the investigational product (IP).
Groups:
- Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL: Participants with R/R solid tumors known to express NY-ESO-1 received IV infusion of ASP0739 (HEK293 transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^7 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a PR or SD (1 cycle= 28 days).
- Total: Total of all reporting groups
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL | Total
Number analyzed (Participants) | 4 | 7 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (3.9) | 50 (14.6) | 46.4 (18.9) | 44.7 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 2 | 4 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 0 | 5
  Not Hispanic or Latino | 0 | 5 | 5 | 10
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 6 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Number of participants with Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Scale was used to assess performance status. Grades: 0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory, able to carry out work of light nature. 2: Ambulatory, capable of self-care, unable to carry out work activities. Up and about more than 50% waking hours. 3: Capable of limited self-care, confined to bed/chair more than 50% waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair. 5: Dead. Only participants with ECOG grades were reported.
  Participants
    Grade 0 | 3 | 4 | 2 | 9
    Grade 1 | 0 | 2 | 3 | 5
    Grade 2 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any event occurring within 28 days of first dose on C1D1 and graded as:
  * Grade (GR) ≥2 autoimmune reaction
  * GR 3 Immune related AEs (irAEs) that did not resolve to GR ≤1 in 3 to 5 days, febrile neutropenia with or without infection, thrombocytopenia with bleeding requiring transfusion, anemia requiring transfusion
  * GR 4 irAEs, neutropenia, thrombocytopenia, anemia
  * GR ≥3 non-hematological AE that did not resolve to GR ≤2 within 72 hours of onset, liver function test abnormality lasting ≥7 days Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 × upper limit of normal (ULN; GR≥3) without liver metastases and 8 × ULN in participants with liver metastases, AST or ALT >3 × ULN and total bilirubin (TBL) >2 × ULN (in participants with, Gilbert syndrome: AST or ALT >3 × ULN and direct bilirubin >1.5) (confirmed Hy's Law)
  * GR 5 toxicity, Prolonged delay (>2 weeks) in initiating cycle 2 due to treatment-related toxicity.
Time Frame: Cycle 1 Day 1 (C1D1) up to C1D28
Population: DLT Evaluation Analysis Set (DEAS).The DEAS was defined as all participants in SAF excluding participants who met any of the following criteria:
  * Participant was discovered to have enrolled without fully satisfying eligibility criteria.
  * Participant received less than the planned dose in cycle 1 for reasons other than DLT.
  * Participant had no DLT and withdrew from the study before the end of DLT evaluation period.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 7 | 5
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) & Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An AE was considered "serious" if, it resulted in any of the following outcomes: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly, or birth defect; requires inpatient hospitalization; or leads to prolongation of hospitalization; other medically important events. A treatment-emergent adverse event (TEAE) was defined as an AE observed after the date of first dose until 30 days after the last dose.
Time Frame: From first dose up to 198 days
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 7 | 5
Participants
  TEAEs | 4 | 7 | 5
  SAEs | 1 | 2 | 1

3. Primary Outcome: Number of Participants With ECOG Performance Status at C1D2
Description: The ECOG Scale was used to assess performance status.
  Grade Description:
  0 - Fully active, able to carry on all pre disease performance without restriction.
  1. - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. - Ambulatory and capable of all self-care, but unable to carry out any work activities.
     Up and about more than 50% of waking hours.
  3. - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. -Dead.
Time Frame: At C1D2
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 6 | 5
Participants
  Grade 0 | 3 | 3 | 2
  Grade 1 | 0 | 3 | 3
  Grade 2 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With ECOG Performance Status at C1D8
Description: as for outcome 3
Time Frame: At C1D8
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 7 | 5
Participants
  Grade 0 | 3 | 4 | 2
  Grade 1 | 0 | 2 | 2
  Grade 2 | 1 | 1 | 1
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With ECOG Performance Status at CID15
Description: as for outcome 3
Time Frame: At CID15
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 7 | 4
Participants
  Grade 0 | 3 | 4 | 3
  Grade 1 | 0 | 2 | 1
  Grade 2 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With ECOG Performance Status at CID22
Description: as for outcome 3
Time Frame: At CID22
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 2 | 6 | 4
Participants
  Grade 0 | 2 | 4 | 3
  Grade 1 | 0 | 2 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With ECOG Performance Status at C2D1
Description: as for outcome 3
Time Frame: At C2D1
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 6 | 4
Participants
  Grade 0 | 3 | 4 | 3
  Grade 1 | 0 | 2 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With ECOG Performance Status at C2D2
Description: as for outcome 3
Time Frame: At C2D2
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 3
Participants
  Grade 0 |  |  | 2
  Grade 1 |  |  | 1
  Grade 2 |  |  | 0
  Grade 3 |  |  | 0
  Grade 4 |  |  | 0
  Grade 5 |  |  | 0

9. Primary Outcome: Number of Participants With ECOG Performance Status at C2D8
Description: as for outcome 3
Time Frame: At C2D8
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Grade 0 | 1 | 3 | 3
  Grade 1 | 1 | 1 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With ECOG Performance Status at C2D15
Description: as for outcome 3
Time Frame: At C2D15
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Grade 0 | 2 | 4 | 2
  Grade 1 | 1 | 2 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With ECOG Performance Status at C2D22
Description: as for outcome 3
Time Frame: At C2D22
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 5 | 2
Participants
  Grade 0 | 2 | 3 | 1
  Grade 1 | 1 | 2 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With ECOG Performance Status at C3D1
Description: as for outcome 3
Time Frame: At C3D1
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1
Participants
  Grade 0 | 1 | 2 | 1
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With ECOG Performance Status at C3D8
Description: as for outcome 3
Time Frame: At C3D8
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 0
Participants
  Grade 0 | 1 | 2 |
  Grade 1 | 0 | 0 |
  Grade 2 | 0 | 0 |
  Grade 3 | 0 | 0 |
  Grade 4 | 0 | 0 |
  Grade 5 | 0 | 0 |

14. Primary Outcome: Number of Participants With ECOG Performance Status at C3D15
Description: as for outcome 3
Time Frame: At C3D15
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 2 | 1
Participants
  Grade 0 |  | 2 | 1
  Grade 1 |  | 0 | 0
  Grade 2 |  | 0 | 0
  Grade 3 |  | 0 | 0
  Grade 4 |  | 0 | 0
  Grade 5 |  | 0 | 0

15. Primary Outcome: Number of Participants With ECOG Performance Status at C3D22
Description: as for outcome 3
Time Frame: At C3D22
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 0
Participants
  Grade 0 | 1 | 2 |
  Grade 1 | 0 | 0 |
  Grade 2 | 0 | 0 |
  Grade 3 | 0 | 0 |
  Grade 4 | 0 | 0 |
  Grade 5 | 0 | 0 |

16. Primary Outcome: Number of Participants With ECOG Performance Status at C4D1
Description: as for outcome 3
Time Frame: At C4D1
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1
Participants
  Grade 0 | 1 | 2 | 1
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With ECOG Performance Status at C4D8
Description: as for outcome 3
Time Frame: At C4D8
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 2 | 0
Participants
  Grade 0 |  | 2 |
  Grade 1 |  | 0 |
  Grade 2 |  | 0 |
  Grade 3 |  | 0 |
  Grade 4 |  | 0 |
  Grade 5 |  | 0 |

18. Primary Outcome: Number of Participants With ECOG Performance Status at C4D15
Description: as for outcome 3
Time Frame: At C4D15
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1
Participants
  Grade 0 | 1 | 2 | 1
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With ECOG Performance Status at C4D22
Description: as for outcome 3
Time Frame: At C4D22
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 0 | 0
Participants
  Grade 0 | 1 |  |
  Grade 1 | 0 |  |
  Grade 2 | 0 |  |
  Grade 3 | 0 |  |
  Grade 4 | 0 |  |
  Grade 5 | 0 |  |

20. Primary Outcome: Number of Participants With ECOG Performance Status at C5D1
Description: as for outcome 3
Time Frame: At C5D1
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 0 | 1
Participants
  Grade 0 | 1 |  | 1
  Grade 1 | 0 |  | 0
  Grade 2 | 0 |  | 0
  Grade 3 | 0 |  | 0
  Grade 4 | 0 |  | 0
  Grade 5 | 0 |  | 0

21. Primary Outcome: Number of Participants With ECOG Performance Status at C5D15
Description: as for outcome 3
Time Frame: At C5D15
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 1
Participants
  Grade 0 |  |  | 1
  Grade 1 |  |  | 0
  Grade 2 |  |  | 0
  Grade 3 |  |  | 0
  Grade 4 |  |  | 0
  Grade 5 |  |  | 0

22. Primary Outcome: Number of Participants With ECOG Performance Status at C6D1
Description: as for outcome 3
Time Frame: At C6D1
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 0 | 1
Participants
  Grade 0 | 1 |  | 1
  Grade 1 | 0 |  | 0
  Grade 2 | 0 |  | 0
  Grade 3 | 0 |  | 0
  Grade 4 | 0 |  | 0
  Grade 5 | 0 |  | 0

23. Primary Outcome: Number of Participants With ECOG Performance Status at C6D15
Description: as for outcome 3
Time Frame: At C6D15
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 1
Participants
  Grade 0 |  |  | 1
  Grade 1 |  |  | 0
  Grade 2 |  |  | 0
  Grade 3 |  |  | 0
  Grade 4 |  |  | 0
  Grade 5 |  |  | 0

24. Primary Outcome: Number of Participants With ECOG Performance Status at End of Treatment (EOT) Visit
Description: The ECOG Scale was used to assess performance status.
  Grade Description:
  0 - Fully active, able to carry on all pre disease performance without restriction.
  1. - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. - Ambulatory and capable of all self-care, but unable to carry out any work activities.
     Up and about more than 50% of waking hours.
  3. - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. -Dead. EOT visit was 7 days after last dose.
Time Frame: At EOT visit (day 175)
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 2 | 7 | 3
Participants
  Grade 0 | 1 | 5 | 2
  Grade 1 | 1 | 1 | 1
  Grade 2 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

25. Primary Outcome: Number of Participants With ECOG Performance Status at Safety Follow up 30 Days
Description: as for outcome 3
Time Frame: At 30 days safety follow up (day 198)
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 1 | 1
Participants
  Grade 0 |  | 1 | 1
  Grade 1 |  | 0 | 0
  Grade 2 |  | 0 | 0
  Grade 3 |  | 0 | 0
  Grade 4 |  | 0 | 0
  Grade 5 |  | 0 | 0

26. Primary Outcome: Number of Participants With ECOG Performance Status at Safety Follow up 60 Days
Description: as for outcome 3
Time Frame: At 60 days safety follow up (day 228)
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Grade 0 | 1 | 1 |
  Grade 1 | 0 | 0 |
  Grade 2 | 0 | 0 |
  Grade 3 | 0 | 0 |
  Grade 4 | 0 | 0 |
  Grade 5 | 0 | 0 |

27. Primary Outcome: Number of Participants With ECOG Performance Status at Safety Follow up 90 Days
Description: as for outcome 3
Time Frame: At 90 days safety follow up (day 258)
Population: SAF with available data analyzed.
Measure: Number; unit: Participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 0 | 0
Participants
  Grade 0 | 1 |  |
  Grade 1 | 0 |  |
  Grade 2 | 0 |  |
  Grade 3 | 0 |  |
  Grade 4 | 0 |  |
  Grade 5 | 0 |  |

28. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The dose recommended for use in phase 2 studies was analyzed on the basis of the safety, tolerability, and preliminary pharmacokinetic (PK) and efficacy data obtained in phase 1 studies.
Time Frame: C1D1 up to C1D28
Population: SAF
Measure: Number; unit: cells/mL
Groups:
- All Participants (Phase 1): Participants with R/R solid tumors known to express NY-ESO-1 received IV infusion of ASP0739 (HEK293 transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^7 cells/mL or 1x10^8 cells/mL; at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a PR or SD (1 cycle= 28 days).
Arm/Group | All Participants (Phase 1)
Number analyzed (Participants) | 11
cells/mL | 1*10^8

29. Primary Outcome: Objective Response Rate Per Immune Response Evaluation Criteria in Solid Tumors (iRECIST) (iORR) by Independent Central Review
Description: iORR was defined as the percentage of participants for each dose level whose best overall response is rated as complete response (iCR) or partial response (iPR) per iRECIST. iORR assessments included:
  * iORR with confirmed response
  * iORR with unconfirmed response
  iCR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: From first dose up to 525 days
Population: Due to early termination of the study, sponsor decided not to collect data for endpoints that were assessed by independent central review, thus data was not reported.
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Objective Response Rate Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (ORR) by Investigator Assessment
Description: ORR was defined as the percentage of participants for each dose level whose best overall response is rated as CR or PR per RECIST v1.1. ORR assessment included:
  ORR with confirmed response ORR with unconfirmed response
  Participants who had CR or PR were considered to have confirmed response, and participants who did not meet this criterion were considered to have unconfirmed response.
  CR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: From first dose up to 525 days
Population: Response Analysis Set (RAS): The response analysis consisted of all participants who were enrolled and received at least one dose of IP and had at least one post baseline primary efficacy measurement.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 6 | 4
Percentage of participants
  Confirmed response | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2]
  Unconfirmed response | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2]

31. Secondary Outcome: Disease Control Rate Per iRECIST (iDCR) by Investigator Assessment
Description: iDCR was defined as the percentage of participants for each dose level whose best overall response is rated as confirmed and unconfirmed iCR, iPR or stable disease (iSD) per iRECIST.
  iCR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 mm in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. SD was defined as neither sufficient shrinkage to qualify for iPR nor sufficient increase to qualify for progressive disease.
  Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
  Participants who had CR or PR were considered to have confirmed response, and participants who did not meet this criterion were considered to have unconfirmed response.
Time Frame: From first dose up to 525 days
Population: RAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 6 | 4
Percentage of participants
  Confirmed response | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9] | 25.0 [0.6 to 80.6]
  Unconfirmed response | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9] | 25.0 [0.6 to 80.6]

32. Secondary Outcome: Disease Control Rate Per RECIST v1.1 (DCR) by Investigator Assessment
Description: DCR is defined as the percentage of participants for each dose level whose best overall response is rated as confirmed CR, PR or SD per RECIST v1.1.CR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 mm in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
  Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: From first dose up to 525 days
Population: RAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 6 | 4
Percentage of participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9] | 25.0 [0.6 to 80.6]

33. Secondary Outcome: Progression-Free Survival Per iRECIST (iPFS) by Independent Central Review
Description: iPFS is defined as the time from the date of first dose until death from any cause or radiographic disease progression assessed per iRECIST by independent central review.
  Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: From first dose up to 525 days
Population: as for outcome 29
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0

34. Secondary Outcome: iPFS Per iRECIST by Investigator Assessment
Description: iPFS is defined as the time from the date of first dose until death from any cause or radiographic disease progression assessed per iRECIST by investigator assessment.
  Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: From first dose up to 525 days
Population: FAS with available data analyzed. The dose level utilized during the expansion phase was the recommended phase 2 dose (RP2D), which was carefully selected from the dose escalation phase and a pooled population was used to estimate time-to-event efficacy endpoints for a comprehensive overview of the treatment's effectiveness
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Dose Escalation and Expansion Phase: ASP0739 1x10^8 Cells/mL: Participants with R/R solid tumors known to express NY-ESO-1 or SS, MRCL, ovarian cancer and other solid tumors known to express NY-ESO-1 (melanoma, NSCLC adenocarcinoma and squamous cell and ESCC) received IV infusion of ASP0739 (HEK293 transfected with a lentiviral vector that is encoding the target antigen NY-ESO-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for a total of 4 doses; an additional 2 doses was administered in participants with a PR or SD (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation and Expansion Phase: ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 10
Days | 81.0 [51.0 to NA] — Due to low number of events, upper limit of 95% CI was not estimable. | 52.5 [43.0 to 106.0]

35. Secondary Outcome: Progression-Free Survival Per RECIST v1.1 (PFS) by Investigator Assessment
Description: PFS is defined as the time from the date of first dose until death from any cause or radiographic disease progression assessed per RECIST v1.1 by investigator assessment.Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started
Time Frame: From first dose up to 525 days
Population: FAS with available data analyzed. The dose level utilized during the expansion phase was the RP2D, which was carefully selected from the dose escalation phase and a pooled population was used to estimate time-to-event efficacy endpoints for a comprehensive overview of the treatment's effectiveness.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation and Expansion Phase: ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 10
Days | 52.0 [51.0 to NA] — Due to low number of events, upper limit of 95% CI was not estimable. | 52.5 [43.0 to 106.0]

36. Secondary Outcome: Duration of Overall Survival (OS)
Description: OS is defined as the time from the date of first dose until the date of death from any cause (death date - first dose date + 1). For a participant who is not known to have died by the end of study follow-up, OS is censored at the date of last contact (date of last contact - first dose date + 1).
Time Frame: From first dose up to 525 days
Population: FAS. The dose level utilized during the expansion phase was the RP2D, which was carefully selected from the dose escalation phase and a pooled population was used to estimate time-to-event efficacy endpoints for a comprehensive overview of the treatment's effectiveness.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation and Expansion Phase: ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 12
Days | 189.5 [10.0 to NA] — Due to low number of events, upper limit of 95% CI was not estimable. | NA [54.0 to NA] — Due to low number of events, median and upper limit of 95% CI was not estimable.

37. Secondary Outcome: Duration of Response Per iRECIST (iDOR)
Description: iDOR as per iRECIST was defined as the time from the date of the first response iCR/iPR (whichever is first recorded) to the date of radiographical progression or date of censoring. iCR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 mm in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: From first response up to 525 days
Population: Due to early termination of the study, sponsor decided not to collect data for this endpoint, thus data was not reported.
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Duration of Response Per RECIST (DOR) v1.1
Description: DOR as per RECIST 1.1 was defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression or date of censoring.
  CR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 mm in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: From first response up to 525 days
Population: as for outcome 37
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0

39. Secondary Outcome: ORR Per iRECIST (iORR) by Investigator Assessment
Description: iORR was defined as the percentage of participants for each dose level whose best overall response is rated as iCR or iPR per iRECIST. iORR assessments included:
  * iORR with confirmed response
  * iORR with unconfirmed response
  iCR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 mm in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
  Participants who had CR or PR were considered to have confirmed response, and participants who did not meet this criterion were considered to have unconfirmed response.
Time Frame: From first dose up to 525 days
Population: RAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 6 | 4
Percentage of participants
  Confirmed response | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2]
  Unconfirmed response | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2]

ADVERSE EVENTS:
Time Frame: For AEs: From first dose up to 198 days. For All-cause mortality: From first dose up to 525 days
Description: SAF. First dose took place at the same time as randomization.
Arm/Group | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/7 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/7 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL (N=4) | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL (N=7) | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL (N=5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation (Phase 1): ASP0739 1x10^7 Cells/mL (N=4) | Dose Escalation (Phase 1): ASP0739 1x10^8 Cells/mL (N=7) | Dose Expansion (Phase 2): ASP0739 1x10^8 Cells/mL (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04939701/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT04939701/SAP_002.pdf